CLINICAL TRIAL: NCT06403189
Title: Profound Cerebral Folate Deficiency as a Clinical Model for Identification of MRI and Biochemical Signatures of Choroid Plexus Dysfunction
Brief Title: Choroid Plexus Dysfunction in Neurological Diseases
Acronym: PLEXFOLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240013
Record Dates: First submitted 2024-04-25; First posted 2024-05-07 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Plexus Choroideus; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: * consultation with a neurologist
  * Biologic samples (blood and lombar punction)
  * MRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Population (Other): * LHIPFOLD patients
  * Patients with neurologic disease
  * healthy volunteers
  Interventions: Other: Biologic samples and MRI

INTERVENTIONS:
Other: Biologic samples and MRI — * blood sample
  * lumbar punction
  * MRI

SUMMARY:
Cerebral folate deficiency (CFD), a partially treatable condition defined by a low folate cerebrospinal fluid (CSF) concentration, can be linked to genetic defects of folate metabolism or be secondary to various diseases without clear causal link. The team identified a neurological syndrome (named LHIPFOLFD) characterized by deep CFD and a specific leukoencephalopathy, related to several possible gene defects never involving folate metabolism. The team hypothesize that CFD in LHIPFOLD is due to a Choroid Plexus (CP) dysfunction, a brain organ that expresses transporters regulating flux between blood and CSF of numerous metabolites (including folate), and secretes CSF and specific proteins. Consequently, other potentially treatable biochemical abnormalities due to PC dysfunction may exist in LHIPFOLD, beyond CFD. Currently, there is no available clinical explorations to evaluate CP functions, whereas the team consider LHIPFOLD a very useful model to validate the capacity of some relevant diagnostic tools to do so. The objectives are to identify a CP-related MRI and biochemical signature in LHIPFOLD patients, using morphological and functional imaging (CP capillary permeability and CP macrovascular perfusion), and metabolomics/proteomics approaches (untargeted then targeted validation of candidate biomarkers related to CP physiology); and to set-up imaging and biochemical diagnostic tests for clinical practice. For this, brain MRI data and blood/CSF samples will be collected during 2 years from LHIPFOLD patients and controls. Some experimental data indicate that the innovative concept of generalized PC dysfunction as part of a more global pathophysiology has the potential to be applied to other neurological diseases like Alzheimer's disease. Therefore, efficient diagnostic tools exploring CP function will be of great utility not only in LHIPFOLD but also in more common neurological diseases, potentially leading to original therapeutic approaches.

DETAILED DESCRIPTION:
Cerebral folate deficiency (CFD) is a condition defined by low concentration (<41 nM) of 5-methyltetrahydrofolate (5MTHF, the biologically active form of folate) in the cerebrospinal fluid (CSF) 1. CFD is considered to be of "primary" origin if it is associated with several genetic diseases involving folate metabolism, leading to severe motor and cognitive manifestations. CFD can also be "secondary", i.e. associated with various definite diseases such as genetic mitochondrial diseases and also unidentified diseases. In secondary CFD, the cause of CFD is not understood. In the center, the team identified 16 CFD patients with common characteristics: deep secondary CFD (5MTHF<10nM whereas blood folate is normal), high protein CSF >1g/L (N<0.5), and a specific involvement of brain white matter, hyperintense on T2-weighted MRI. The team called this syndrome "LHIPFOLD" for Leukoencephalopathy with CSF HIgh Protein and FOLate Deficiency (confidential, planned submission in end of 2022). Within the French metabolic biochemistry labs network, the team identified 6 additional LHIPFOLDpat (LHIPFOLD patients). They have a mean age of 42 to 14 years (min 15; max 77), and a sex ratio of 1.8 (M/F). 9/22 had either a large mitochondrial DNA deletion (Kearns-Sayre) or bi-allelic POLG mutations (mitochondrial DNA replication defect). The other 13 patients were all undiagnosed until recently, but the team found in a research context and validated in vitro bi-allelic variants in 4/7 tested patients within genes from MRPS family, coding for sub-units of the mitoribosome.

LHIPFOLD patients clearly have a defect of intracerebral 5MTHF transport, but without mutation of the brain folate transporters. Since folate is exclusively transported from blood to the brain by the choroid plexus (CP)2, the team hypothesize that CFD in LHIPFOLD is due to CP dysfunction. CP, localized in the brain ventricles, is a vascularized epithelial organ that acts as a blood-CSF barrier, expressing numerous transporters for molecules transfer from the blood to the CSF and vice versa (removing waste products from brain cells). CP also secretes CSF and expresses CSF-secreted proteins related to various functions3.

High protein CSF due to a blood brain barrier alteration, and reported abnormal CP morphology from brain autopsy in two Kearns-Sayre patients are also in favor of CP dysfunction in LHIPFOLD 4. In addition, in two LHIPFOLDpat, the team found very high concentrations of CSF sialic acid without the involvement of sialic acid-related genes whereas CP strongly expresses the sialic acid efflux transporter. The team also recently measured strongly decreased CP size after automatic segmentation in two other LHIPFOLD pat. All these data strongly argue for CP dysfunction in LHIPFOLD .

If the hypothesis is correct, it means that beyond CFD, other CSF abnormalities probably exist as a consequence of generalized CP dysfunction. This may be very interesting in terms of therapeutic approach, as folate supplementation has a clear but limited therapeutic effect, especially in some patients. Unfortunately, to assess our hypothesis, there is no available clinical exploration to evaluate CP functions, whereas CP dysfunction/alteration is suggested as a potential pathogenesis contributor in several common neurological diseases (for the following text the team will use dysfunction for both dysfunction and alteration). As the team think that in LHIPFOLD the CP dysfunction is particularly severe, as suggested by the deep CFD, the team consider LHIPFOLD syndrome a very useful clinical model to validate the capacity of some relevant diagnostic tools to evaluate CP function. Therefore, the objectives of the project are:

1. Prove CP dysfunction in LHIPFOLD, through the identification of specific and CP-related MRI and biochemical signatures, using CP-centered imaging and metabolomics and proteomics approaches.
2. Identify CP-related biochemical biomarkers in LHIPFOLD directly amenable to treatment.
3. Set-up imaging and biochemical diagnostic tests for evaluating CP function in clinical practice (biomarkers-based CP-dysfunction score).

Methodology To reach the objectives, the team will conduct a monocentric diagnostic phase 1 case-control study, based on descriptive, deterministic statistic and multidimensional clustering approach, supported by complementary diagnostic tools specifically designed for CP exploration of LHIPFOLDpat versus healthy volunteers (HV) and neurological control patients (NCpat). NCpat will be used to assess the specificity of the CP-related signatures identified in LHIPFOLDpat. The team expect that findings will be similar to HV in some NCpat, but will reflect slight to moderate CP dysfunction in others. With AP-HP as the study sponsor, the team will obtain approval of the Research Ethics Committee for a "Jardé 1" study, in accordance with the legislation and regulatory requirements in force.

-Patients and controls selection and recruitment Subjects will be prospectively recruited during a two-year period: 1)LHIPFOLDpat will be selected as previously described; 2)HV will be recruited by the usual advertisement procedure, and will be matched for age and sex with LHIPFOLDpat; 3) NCpat will be age and sex matched patients with definite common brain diseases frequently explored in the Neurology department: multiple sclerosis, amyotrophic lateral sclerosis, alzheimer's disease, frontotemporal dementia, idiopathic intracranial hypertension and normal pressure hydrocephalus. The diagnosis of these diseases will be made according to the newest guidelines by the neurologists specialised in each disease. Concerning the sample to be recruited, the team took into account two constraints: the number of LHIPFOLDpat is limited; the study is not a simple deterministic comparison vs a control group but more a multidimensional analysis leading to the identification of CP-related signatures through homogeneous patient clusters. Consequently, the strategy was to identify a global sample size that would lead to a homogeneous classification of patients based on 5 or 6 biomarkers. According to Donicar's formula5 2^6 patients properly selected by a stratified sampling technique should allow this. These 64 patients will include 15 LHIPFOLDpat and an equal number of 25 HV and 25 NCpat. Furthermore, keeping the deterministic approach, and based on a simulation study integrating mean and standard deviation of CSF 5MTHF in LHIPFOLDpat and NCpat (3.85 +/- 2.67 and 49.53 +/- 13.35 respectively) with respectively 15 and 25 subjects, this sample size provides a power greater than 95% to demonstrate a difference with a Wilcoxon Rank Sum test between these two groups (of note, values in HV are currently unknown).

The team will acquire brain MRI data (with blood gadolinium injection), blood and CSF samples from all subjects. LHIPFOLDpat and NCpat will undergo these procedures as part of standard care in the Neurology Department of Pitié-Salpêtrière Hospital. HV will be hospitalized one day in our Clinical Investigation Center. All subjects will sign informed consent and agree to undergo MRI examination and blood and CSF sampling for research purpose for HV, and additional MRI time acquisition and sample volumes for patients.

* Brain MRI study Brain MRI will be performed at 3 TESLA (Siemens PRISMA) at the Centre for Neuroimaging Research (CENIR), the imaging platform of the Paris Brain Institute (ICM). The team will assess both CP morphology and function: 1/for CP morphological analysis, the team will measure CP volumes and extract textural parameters. CP segmentation will be performed using automated software developed at the site. Texture analysis will be performed using the MP2RAGE MRI sequence. 2/CP function assessment will include quantitative measurements of the capillary permeability and macrovascular perfusion. To explore CP permeability, dynamic T1 perfusion sequence with gadolinium enhancement will be used; t-TRANS and other regional values will be extracted. Post processing will be performed using Syngovia (Siemens) software. To explore CP macrovascular perfusion, the team will use a shorter version of the dynamic Arterial Spin Labeling perfusion (without gadolinium) published previously 6. With this sequence the team will be able to appreciate the arterial transit time and apparent blood flow. Data analysis will be performed at CENIR.
* Discovery of CP dysfunction biomarker candidates in CSF/blood compartments Two mixed approaches will be used to select the top 10 biomarkers candidates (a priori 5 metabolites and 5 proteins) that will be investigated by a targeted and fully quantitative analysis: i)untargeted metabolomics and proteomics (the findings will be reviewed to assess a possible link with CP function); and ii)hypothesis-driven approach: in addition to 5MTHF, based on data from the literature and publicly available biological database, the team also identified metabolites (including ascorbic acid and sialic acid) that seem to be specifically transported by the CP, and proteins specifically expressed by the CP (including TRPM3 and Klotho). As blood concentrations can influence CSF concentrations for some molecules, the team plan to analyze blood and CSF sampled at the same time, with calculation of a CSF/Blood ratio of concentrations.

For untargeted metabolomics, metabolic extracts of CSF and plasma samples will be obtained following methanol-assisted protein precipitation and analysed by liquid chromatography coupled to high resolution mass spectrometry (LC-HRMS) as the team routinely perform 7. A combination of two complementary LC-HRMS platforms will be used to profile both hydrophobic and polar metabolites8. Data pre-treatment and statistical analyses will be achieved by using Workflow4Metabolomics (W4M), which is an open-source collaborative online platform for computational metabolomics. Annotation of data sets and identification of biologically relevant signals will be performed by using 'in-house' spectral libraries, and MS/MS (tandem mass spectrometry) experiments. Relative quantification of ~250 metabolites will be achieved thanks to normalization using quality control samples. For targeted metabolomics, CSF 5MTHF is routinely measured in Necker laboratory specialized in Neurometabolism, using very sensitive and specific analytical methods (liquid chromatography hyphenated to tandem MS). The team are in the process to include in the same run ascorbic acid and sialic acid measures. Depending on the chemical nature of the metabolite biomarker candidates identified in the untargeted study, one or few new methods for robust quantification using stable isotopes will be developed.

A preliminary proteomic study on the CSF of a patient with high CSF protein and a control will allow us to establish a sample preparation protocol, select a mass spectrometry analysis method and data analyses workflow. The objective is twofold: to optimize the extraction of proteins and to allow the comparison of very different CSFs in order to develop an analytical strategy that will allow us to identify biomarkers. The study will be carried out by using a label-free approach to minimize variability, the number of steps and especially not to restrict the dynamic range of the sample. All bioinformatics analyses will be performed with myProMS9, our proteomic data management and analysis software developed at the Institut Curie in collaboration with the INSERM U900 bioinformatics platform directed by Dr E. Barillot. For the targeted proteomic approach, the team will use the expertise on targeted MS with stable isotope-labeled internal standard peptides, the gold standard approach for protein quantification in biological fluid, resulting in high robustness, high sensitivity and multiplex analysis10.

-Cross data analysis The team will centrally manage, analyze and integrate clinical and biological datasets and knowledge generated by the MRI and biological samples analysis to identify a global CP-related signature in LHIPFOLD patients. With these data, the team will establish a CP-dysfunction score for use in routine clinical practice, intended to be used to explore CP in neurological patients.

ELIGIBILITY:
Inclusion Criteria:

For LHIPFOLD patients:

* Suspicion of diagnosis or diagnosis of LHIPFOLD syndrome documented in the medical record, i.e. presence of these three manifestations: severe intrathecal deficiency in 5MTHF< 10 nmol/L, hyperproteinorachia > 1 g/L, and white matter abnormalities on cerebral MRI.
* Patient covered by Social Security or Complementary Health Insurance or any equivalent scheme (including AME).

For Neurological Controls (NC) :

* No chronic pathology (notably no renal, cardiac, pulmonary or hepatic disease)
* Patients with one of the following neurological pathologies (confirmed diagnosis or strong suspicion), investigated in the course of routine clinical practice: Alzheimer's disease, multiple sclerosis, amyotrophic lateral sclerosis, intracranial hypertension, normal pressure hydrocephalus, frontotemporal dementia.

For Healthy Volunteers (VS):

* No chronic pathology (in particular, no renal, cardiac, pulmonary, hepatic or psychiatric disease)
* No history of neurological pathology
* No chronic alcohol intoxication
* No consumption of toxic substances in the week preceding the inclusion visit
* No neurological or psychotropic medication.

Exclusion Criteria:

For all research participants:

* Age <18
* Pregnant and breast-feeding women.
* Participant unable to give informed consent.
* Participant with a contraindication to MRI: implantable cardiac defibrillators, prostheses, transdermal patches, catheters; implantable pumps; artificial heart valves; implants to treat deafness (if incompatible with MRI); surgical neurostimulator clips., pregnancy, extreme claustrophobia.
* Participants with contraindications to contrast injection: known allergy to gadolinium chelates, moderate or severe renal insufficiency, pregnancy (BHCG for women of childbearing age prior to MRI), breast-feeding.
* Participants with contraindications to LP: haemostasis abnormalities (PT<50%, platelets < 40*109/L), mass syndrome on brain imaging, suspected infection at or near the needle insertion site, coagulopathy, cardiopulmonary insufficiency or respiratory distress.

For NC and VS :

* Participant under legal protection (guardianship, curatorship)
* Participant not covered by Social Security or Complementary Health Insurance or any equivalent scheme (excluding AME).
* Taking folate, vitamin C or dietary supplements containing vitamins in the two months prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2028-02-03 (Estimated); Study Completion 2028-02-03 (Estimated)

PRIMARY OUTCOMES:
Identify a clinico-radio-proteo-metabolic profile indicative of choroid plexus dysfunction based on observation of LHIPFOLD patients as an experimental model. | 37 months
  Characterization of a specific combined biochemical and radiological signature associated with choroid plexus damage observed in LHIPFOLD patients considered as "cases", comprising a limited number of biomarkers (target 5 to 6).

SECONDARY OUTCOMES:
Development of a simple diagnostic strategy based on biochemistry (metabolites/proteins) of blood and CSF discriminating choroid plexus alteration, using LHIPFOLD patients as an experimental model. | 37 months
  Development of a biochemical diagnostic kit (proteins and metabolites) discriminating (sensitive and specific) PC dysfunction. The proposed analytical approach will be built as a back-and-forth between analyses carried out within the framework of the main objective on metadata and analyses carried out by data category. Still taking the point of view of a data-driven analysis and using supervised and unsupervised learning methods, the aim here will be to define different classifiers: a global classifier and thematic classifiers (1 for proteins, 1 for metabolites) that will perform well in classifying PC dysfunctions. These classifiers could be used to develop diagnostic kits for routine use.
Development of a simple MRI diagnostic strategy (acquisition and analysis) that can be used routinely for the radiological identification of choroid plexus damage, based on the observation of LHIPFOLD patients as an experimental model. | 37 months
  Set up an MRI acquisition and image analysis protocol that is sensitive and specific to PC dysfunction.
Identification of therapeutic targets, i.e. blood and CSF biochemical biomarkers indicating choroid plexus dysfunction AND likely to be modulated by therapeutic intervention (e.g. supplementation of DFIC with folinic acid). | 37 months
  In order to identify potential therapeutic targets, a network-based biologic analysis will be carried out. The expected deliverables for this objective are the production of biological interaction networks and the identification of one or more therapeutic targets. The measurable evaluation criteria are represented here by the centrality indices of the various biomarkers identified within the biological networks. The aim of this analysis will be to identify the proteins or metabolites with the most central role in the network, and for which variations would produce the greatest impact on the biological network as a whole, and thus provide priority therapeutic targets.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CIC Neurosciences, Paris
  - Service de Neurologie, Pitié-Salpêtrière, Paris